CLINICAL TRIAL: NCT06360081
Title: Bioequivalence of Zongertinib Tablets From Two Different Manufacturers Following Oral Administration in Healthy Male and Female Subjects (an Open-label, Randomised, Single-dose, Two-period, Two-sequence Crossover Trial)
Brief Title: A Study in Healthy People to See How Zongertinib is Taken up Into the Blood When Given as Tablets Made by Two Different Manufacturers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1479-0019; 2023-510495-31-00 (Other: CTIS); U1111-1303-4345 (Other: WHO)
Record Dates: First submitted 2024-04-08; First posted 2024-04-11 (Actual); Results first posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Zongertinib (manufacturer 1) Test followed by zongertinb (manufacturer 2) Reference treatment (T-R) (Experimental): Participants were administered during Period 1 on Day 1 a single oral dose of 60 milligrams (mg) of zongertinib film-coated tablet produced by Manufacturer 1 (Test treatment, T) with 240 milliliters (ml) of water following an overnight fast of at least 10 hours (hrs). Following a washout period of at least 14 days, participants were administered a single oral dose of 60 mg of zongertinib produced by Manufacturer 2 (Reference treatment, R) with 240 mL of water after an overnight fast of at least 10 hrs.
  Interventions: Drug: Zongertinib manufacturer 1; Drug: Zongertinib manufacturer 2
- Zongertinib (manufacturer 2) Reference followed by zongertinb (manufacturer 1) Test treatment (R-T) (Experimental): Participants were administered during Period 1 on Day 1 a single oral dose of 60 mg of zongertinib film-coated tablet produced by Manufacturer 2 (Reference treatment, R) with 240 ml of water following an overnight fast of at least 10 hrs. Following a washout period of at least 14 days, participants were administered a single oral dose of 60 mg of zongertinib produced by Manufacturer 1 (Test treatment, T) with 240 mL of water after an overnight fast of at least 10 hrs.
  Interventions: Drug: Zongertinib manufacturer 1; Drug: Zongertinib manufacturer 2

INTERVENTIONS:
Drug: Zongertinib manufacturer 1 — Zongertinib
  Other Names: BI 1810631, Hernexeos®
Drug: Zongertinib manufacturer 2 — Zongertinib
  Other Names: BI 1810631, Hernexeos®

SUMMARY:
The main objective of this trial is to establish the bioequivalence of zongertinib tablet from manufacturer 1 (Test, T) compared with zongertinib tablet from manufacturer 2 (reference, R) following oral administration.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (blood pressure (BP), pulse rate (PR)), 12-lead electrocardiogram (ECG), and clinical laboratory tests
* Age of 18 to 50 years (inclusive)
* BMI (Body mass index) of 18.5 to 29.9 kg/m2 (inclusive)
* Signed and dated written informed consent in accordance with ICH-GCP and local legislation prior to admission to the trial
* Either male subject, or female subject who meet any of the following criteria for a highly effective contraception from at least 30 days before the first administration of trial medication until 30 days after trial completion:

  * Use of progestogen-only hormonal contraception that inhibits ovulation (only injectables or implants), plus condom
  * Use of intrauterine device (IUD) or intrauterine hormone-releasing system (IUS)
  * Sexually abstinent
  * A vasectomised sexual partner who received medical assessment of the surgical success (documented absence of sperm) and provided that partner is the sole sexual partner of the trial participant
  * Surgically sterilised (including hysterectomy or bilateral tubular occlusion)
  * Postmenopausal, defined as no menses for 1 year without an alternative medical cause (in questionable cases a blood sample with levels of follicle stimulating hormone (FSH) above 40 U/L and estradiol below 30 ng/L is confirmatory)

Exclusion Criteria:

* Any finding in the medical examination (including BP, PR or ECG) deviating from normal and assessed as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 50 to 90 bpm
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease assessed as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy or simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts Further exclusion criteria apply.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2024-04-30 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-07-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- CRS Clinical Research Services Mannheim GmbH, Mannheim, Germany

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to:
  https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an open-label, randomised, single-dose, two-period and two-sequence crossover trial in healthy male and female subjects to compare a test treatment (T) to a reference treatment (R). The test and reference treatments comprised 60 mg zongertinib tablet manufactured by two different manufacturers.
  Subjects were randomly allocated to the two treatment sequences, namely T-R or R-T (i.e. all subjects received both treatments), with a washout period of at least 14 days between treatments.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Groups:
- First Zongertinib Test, Then Zongertinib Reference (T-R): Participants were administered during Period 1 on Day 1 a single oral dose of 60 milligrams (mg) of zongertinib film-coated tablet produced by Manufacturer 1 (Test treatment, T) with 240 milliliters (ml) of water following an overnight fast of at least 10 hours (hrs).
  Following a washout period of at least 14 days, participants were administered a single oral dose of 60 mg of zongertinib produced by Manufacturer 2 (Reference treatment, R) with 240 mL of water after an overnight fast of at least 10 hrs.
- First Zongertinib Reference, Then Zongertinib Test (R-T): Participants were administered during Period 1 on Day 1 a single oral dose of 60 mg of zongertinib film-coated tablet produced by Manufacturer 2 (Reference treatment, R) with 240 ml of water following an overnight fast of at least 10 hrs.
  Following a washout period of at least 14 days, participants were administered a single oral dose of 60 mg of zongertinib produced by Manufacturer 1 (Test treatment, T) with 240 mL of water after an overnight fast of at least 10 hrs.
Period: Treatment Period 1 (Day 1)
Arm/Group | First Zongertinib Test, Then Zongertinib Reference (T-R) | First Zongertinib Reference, Then Zongertinib Test (R-T)
Started | 28 | 28
Completed | 28 | 28
Not Completed | 0 | 0
Period: Washout Period (14 Days)
Arm/Group | First Zongertinib Test, Then Zongertinib Reference (T-R) | First Zongertinib Reference, Then Zongertinib Test (R-T)
Started | 28 | 28
Completed | 28 | 28
Not Completed | 0 | 0
Period: Treatment Period 2
Arm/Group | First Zongertinib Test, Then Zongertinib Reference (T-R) | First Zongertinib Reference, Then Zongertinib Test (R-T)
Started | 28 | 28
Completed | 28 | 28
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS): The treated set included all subjects who were treated with at least one dose of the trial drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | First Zongertinib Test, Then Zongertinib Reference (T-R) | First Zongertinib Reference, Then Zongertinib Test (R-T) | Total
Number analyzed (Participants) | 28 | 28 | 56
Age, Continuous [Mean (Standard Deviation); unit: Years] | 32.5 (9.0) | 31.7 (7.7) | 32.1 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 10 | 18
  Male | 20 | 18 | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 27 | 27 | 54
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 27 | 26 | 53
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve of Zongertinib in Plasma Over the Time Interval From 0 to 72h (AUC0-72h)
Description: Area under the concentration-time curve of zongertinib in plasma over the time interval from 0 to 72h (AUC0-72h) is reported. Geometric least squares mean (adjusted geometric mean) and adjusted geometric standard error were calculated using an analysis of variance model (ANOVA) on the logarithmic scale. The pharmacokinetic (PK) endpoints were log-transformed (natural logarithm) prior to fitting the ANOVA model. The model included 'subjects within sequences' as a random effect, and sequence, period and treatment as fixed. These quantities were then back transformed to the original scale to provide the point estimate and 90% confidence intervals (CIs) for each endpoint.
Time Frame: Within 3 hours prior to and 0.50, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 10, 12, 24, 36, 48, and 72 hours after administration of zongertinib Test Treatment and zongertinib Reference Treatment.
Population: Pharmacokinetic (PK) parameter analysis set (PKS): This set included all subjects in the treated set (TS) who provided at least 1 primary or secondary PK endpoint and were not excluded due to a protocol deviation relevant to the evaluation of PK or due to PK non-evaluability.
Measure: Geometric Least Squares Mean (Standard Error); unit: hours*nanomole/Liter (h·nmol/L)
Groups:
- Zongertinib Test Treatment (T): This arm included all participants who received a single oral dose of zongertinib tablet (60 mg tablet) produced by Manufacturer 1 (Test Treatment, T).
- Zongertinib Reference Treatment (R): This arm included all participants who received a single oral dose of zongertinib tablet (60 mg tablet) produced by Manufacturer 2 (Reference Treatment, R)
Arm/Group | Zongertinib Test Treatment (T) | Zongertinib Reference Treatment (R)
Number analyzed (Participants) | 56 | 56
hours*nanomole/Liter (h·nmol/L) | 13448.03 (NA) — Adjusted geometric standard error = 1.03 | 13463.07 (NA) — Adjusted geometric standard error = 1.03
Statistical Analysis 1: Comparison: Zongertinib Test Treatment (T) vs Zongertinib Reference Treatment (R); PK endpoints were back transformed to the original scale to provide the point estimate and 90% confidence intervals (CIs) for each endpoint. The model included effects accounting for variation in sequence, subjects within sequences, period, and treatment. The effect 'subjects within sequences' was considered as random, whereas the others were considered as fixed. Confidence intervals were calculated based on the residual error from the ANOVA; Test type: Equivalence — The assessment of bioequivalence was based on two-sided 90% CIs for the ratios of the geometric means (gMean) (T/R) using an acceptance range of 80.0 to 125.0%; p < 0.0001, ANOVA — p-value was calculated for ratios outside the 80.0 to 125.0% interval; Ratio of adjusted geometric means (T/R) = 99.89, 90% CI 2-sided [97.08 to 102.78] — Ratio as percentage [%] Intra-individual geometric coefficient of variation (gCV) = 9.0%

2. Primary Outcome: Maximum Measured Concentration of Zongertinib in Plasma (Cmax)
Description: Maximum measured concentration of zongertinib in plasma (Cmax) is reported. Geometric least squares mean (adjusted geometric mean) and adjusted geometric standard error were calculated using an analysis of variance model (ANOVA) on the logarithmic scale. The pharmacokinetic (PK) endpoints were log-transformed (natural logarithm) prior to fitting the ANOVA model. The model included 'subjects within sequences' as a random effect, and sequence, period and treatment as fixed. These quantities were then back transformed to the original scale to provide the point estimate and 90% confidence intervals (CIs) for each endpoint.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Least Squares Mean (Standard Error); unit: nanomole/Liter (nmol/L)
Arm/Group | Zongertinib Test Treatment (T) | Zongertinib Reference Treatment (R)
Number analyzed (Participants) | 56 | 56
nanomole/Liter (nmol/L) | 1135.49 (NA) — Adjusted geometric standard error = 1.04 | 1126.11 (NA) — Adjusted geometric standard error = 1.04
Statistical Analysis 1: Comparison: Zongertinib Test Treatment (T) vs Zongertinib Reference Treatment (R); [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.0001, ANOVA — p-value was calculated for ratios outside the 80.0 to 125.0% interval; Ratio of adjusted geometric means (T/R) = 100.83, 90% CI 2-sided [96.43 to 105.44] — Ratio as percentage [%] Intra-individual geometric coefficient of variation (gCV) = 14.2%

3. Secondary Outcome: Time From Dosing to Maximum Measured Concentration of Zongertinib in Plasma (Tmax)
Description: Time from dosing to maximum measured concentration of zongertinib in plasma (tmax) is reported.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: hours (h)
Arm/Group | Zongertinib Test Treatment (T) | Zongertinib Reference Treatment (R)
Number analyzed (Participants) | 56 | 56
hours (h) | 2.50 [1.00 to 4.00] | 2.01 [1.00 to 4.03]

ADVERSE EVENTS:
Time Frame: Serious Adverse Events and Other Adverse Events: From study drug administration until end of the residual effect period (i.e. 14 days), up to 336 hours. All-cause mortality: From drug administration till end of trial, up to 18 days.
Description: Treated set (TS): The treated set included all subjects who were treated with at least one dose of the trial drug.
Arm/Group | Zongertinib Test Treatment (T) | Zongertinib Reference Treatment (R)
All-Cause Mortality (participants affected / at risk) | 0/56 | 0/56
Serious Adverse Events (participants affected / at risk) | 0/56 | 0/56
Other Adverse Events (participants affected / at risk) | 13/56 | 13/56
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Zongertinib Test Treatment (T) (N=56) | Zongertinib Reference Treatment (R) (N=56)
Diarrhoea (Gastrointestinal disorders) | 3 | 3
Nausea (Gastrointestinal disorders) | 3 | 2
Fatigue (General disorders) | 5 | 2
Headache (Nervous system disorders) | 8 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2024-03-14): https://cdn.clinicaltrials.gov/large-docs/81/NCT06360081/Prot_000.pdf
  • Statistical Analysis Plan (2024-07-18): https://cdn.clinicaltrials.gov/large-docs/81/NCT06360081/SAP_001.pdf